CLINICAL TRIAL: NCT01147640
Title: A Multicenter, Double-Blind, Randomized, Phase 2 Study to Compare the Safety and Efficacy of Intravenous CXA 101/ Tazobactam and Metronidazole With That of Meropenem in Complicated Intraabdominal Infections
Brief Title: Safety and Efficacy Study to Compare IV CXA 101/Tazobactam and Metronidazole With Meropenem in Complicated Intraabdominal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625A-012; CXA-IAI-10-01 (Other: Cubist Study Number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Complicated Intra-abdominal Infection
MeSH Terms: interventions — ceftolozane; Tazobactam; Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXA 101/tazobactam and metronidazole (Experimental)
  Interventions: Drug: CXA-101/ tazobactam and metronidazole
- meropenem with matching saline placebo (Active Comparator)
  Interventions: Drug: meropenem plus saline placebo

INTERVENTIONS:
Drug: CXA-101/ tazobactam and metronidazole — CXA-101/tazobactam (1000/500 mg q8h) plus metronidazole (500 mg q8h) administered via IV infusion
  Arms: CXA 101/tazobactam and metronidazole
Drug: meropenem plus saline placebo — meropenem IV infusion (1000 mg q8h) plus a matching saline placebo (q8h) administered via IV infusion
  Arms: meropenem with matching saline placebo

SUMMARY:
A Phase 2, multicenter, prospective, randomized, double-blind study of CXA-101/ tazobactam (1000/500 mg q8h) and metronidazole (500 mg q8h) IV infusion vs. meropenem IV infusion (1000 mg q8h) and a matching saline placebo (q8h) in the treatment of cIAI in adult subjects. Dose adjustments for subjects with mild renal impairment are not necessary and subjects with more severe degrees of renal failure are excluded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, from 18 to 90 years of age, inclusive
* One of the following diagnoses (in which there is evidence of intraperitoneal infection) including:(a) Cholecystitis (including gangrenous cholecystitis) with rupture, perforation, or progression of the infection beyond the gallbladder wall;(b)Diverticular disease with perforation or abscess; (c) Appendiceal perforation or periappendiceal abscess; (d) Acute gastric or duodenal perforation, only if operated on >24 hours after perforation occurs; (e) Traumatic perforation of the intestine, only if operated on > 12 hours after perforation occurs; (f) Peritonitis due to perforated viscus, postoperative or spread from other focus of infection (but not spontaneous [primary] bacterial peritonitis or peritonitis associated with cirrhosis and chronic ascites).Subjects with inflammatory bowel disease or ischemic bowel disease are eligible provided there is bowel perforation; or (g) Intraabdominal abscess (including liver and spleen).
* Subject requires surgical intervention (e.g. laparotomy, laparoscopic surgery, or percutaneous draining of an abscess) within 24 hours of (before or after) the first dose of study drug
* If subject is to be enrolled preoperatively, the subject must have radiographic evidence of bowel perforation or intraabdominal abscess
* Subjects who failed prior antibacterial treatment for the current cIAI can be enrolled but must: (a) have a positive culture (from an intraabdominal site) and (b) require surgical intervention. Such subjects can be enrolled before the results of the culture are known; however, if the culture is negative, study drug administration must be discontinued.
* Willing and able to comply with all study procedures and restrictions
* Willing and able to provide written informed consent

Exclusion Criteria:

* Women who are pregnant, nursing, or - if of child bearing potential - not using a medically accepted, effective method of birth control (e.g. condom, oral contraceptive, indwelling intrauterine device, or sexual abstinence)
* Diagnosis of abdominal wall abscess; small bowel obstruction or ischemic bowel disease without perforation; traumatic bowel perforation with surgery within 12 hours; perforation of gastroduodenal ulcer with surgery within 24 hours (these are considered situations of peritoneal soiling before infection has become established); another intraabdominal process in which the primary etiology is not likely to be infectious.
* Simple cholecystitis, gangrenous cholecystitis without rupture, simple appendicitis, acute suppurative cholangitis, infected, necrotizing pancreatitis, or pancreatic abscess
* cIAI managed by staged abdominal repair (STAR), open abdomen technique or any situation where infection source control is not likely to be achieved
* Known prior to randomization to have an IAI or postoperative infection caused by pathogen(s) resistant to meropenem
* Considered unlikely to survive the 4- to 5-week study period
* Any rapidly-progressing disease or immediately life-threatening illness (including acute hepatic failure, respiratory failure and septic shock)
* The need for concomitant systemic antibacterial agents (other than vancomycin or linezolid) in addition to study drug(s)
* Moderate or severe impairment of renal function (estimated CrCl < 50 mL/min), or requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (< 20 mL/h urine output over 24 hours)
* The presence of hepatic disease defined as: (a) ALT or AST > 4 x ULN; (b)Total bilirubin >2 x ULN, unrelated to cholecystitis (c) Alkaline phosphatase >4 x ULN. Subjects with a value >4 x ULN and <5 x ULN are eligible if this value is historically stable.
* Subjects with acute hepatic failure or acute decompensation of chronic hepatic failure
* Hematocrit < 25% or hemoglobin < 8 gm/dL
* Neutropenia with absolute neutrophil count < 1000/mm3
* Platelet count < 75,000 /mm3. Subjects with a platelet count as low as 50,000 /mm3 are permitted if the reduction is historically stable.
* Immunocompromising illness, including known human immunodeficiency virus (HIV) positivity or AIDS, organ (including bone marrow) transplant recipients, and hematological malignancy. Immunosuppressive therapy, including use of high-dose corticosteroid therapy (e.g. >40 mg prednisone or equivalent per day for greater than 2 weeks).
* History of hypersensitivity reactions to cephalosporins, carbapenems, penicillins, ß-lactamase inhibitors, metronidazole, or nitroimidazole derivatives. Subjects with a history of mild skin rash, not documented to be caused by previous ß-lactam use, may be enrolled.
* Any condition or circumstance that, in the opinion of the Investigator, would compromise the safety of the subject or the quality of study data
* Clinically significant abnormality in baseline electrocardiogram (ECG)
* Participation in any investigational drug or device study within 30 days prior to study entry
* Use of systemic antibiotic therapy for IAI for 24 or more hours in the 48-hour period prior to the first dose of study drug, unless there is a documented treatment failure with such therapy
* More than one dose of an active non-study antibacterial regimen was given postoperatively. For subjects enrolled preoperatively, no postoperative non-study antibacterial therapy is allowed
* who previously participated in a study with CXA-101
* Subjects who previously received imipenem, meropenem, doripenem or cefepime for the current intraabdominal infection
* Subjects who have received disulfiram in the past 14 days or who are currently receiving probenecid.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-06-25 (Actual); Primary Completion 2011-02-20 (Actual); Study Completion 2011-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Friedland, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (33):
- United States (11):
  - Pulmonary Consultants and Primary Care Physicians Medical Group, Inc., Orange, California
  - Los Angeles Biomedical Research Institue at Harbor UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Christiana Care Health System, Newark, Delaware
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Metro Health Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Tennessee Health Science Center, Memphis, Tennessee
- Argentina (6):
  - Hospital San Martín, Paraná, Entre Ríos Province
  - Sanatorio Guemes, C.a.b.a.
  - Hospital Nuestra Señora de la Misericordia, Córdoba
  - Hospital San Roque, Córdoba
  - Hospital Central de Mendoza, Mendoza
  - Hospital Dr. José María Cullen, Santa Fe
- Georgia (4):
  - Ltd Ivane Javakhishvili Tbilisi State University Center, Tbilisi
  - JSC K.Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Ltd Vakhtang Bochorishvili Antiseptic Center, Tbilisi
  - Tbilisi State Hospital #4, Tbilisi
- Russia (8):
  - Federal State Institution, Moscow
  - State Moscow Healthcare, Moscow
  - State Healthcare Institution, Moscow
  - Municipal Healthcare Institution "City Clinical Hospital #2", Novosibirsk
  - Regional State Healthcare, Novosibirsk
  - State Healthcare Institution, Saint Petersburg
  - State Educational Institution of Higher Professional Education, Saint Petersburg
  - Saint Petersburg State Healthcare Institution "City Hospital # 26", Saint Petersburg
- Serbia (4):
  - Clinical Hospital Centre Zvezdara, Belgrade
  - Emergency Centre, Clinical Centre of Serbia, Belgrade
  - Clincal Centre Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Lucasti C, Hershberger E, Miller B, Yankelev S, Steenbergen J, Friedland I, Solomkin J. Multicenter, double-blind, randomized, phase II trial to assess the safety and efficacy of ceftolozane-tazobactam plus metronidazole compared with meropenem in adult patients with complicated intra-abdominal infections. Antimicrob Agents Chemother. 2014 Sep;58(9):5350-7. doi: 10.1128/AAC.00049-14. Epub 2014 Jun 30. PMID 24982069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CXA 101/Tazobactam and Metronidazole | Meropenem With Matching Saline Placebo
Started | 83 | 39
Completed | 78 | 38
Not Completed | 5 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Didn't meet eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Microbiological Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | CXA 101/Tazobactam and Metronidazole | Meropenem With Matching Saline Placebo | Total
Number analyzed (Participants) | 82 | 39 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (18.79) | 46.4 (18.48) | 47.8 (18.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 15 | 52
  Male | 45 | 24 | 69

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response of CXA 101/Tazobactam and Metronidazole at Test of Cure (TOC) Visit in the Microbiological Modified Intent to Treat (mMITT) Analysis Population
Description: Clinical response is complete resolution or significant improvement of all signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure was required for the index infection.
Time Frame: Test-of-Cure Visit (7-14 days after End of Therapy [EOT])
Population: mMITT: Treated subjects, with baseline pathogen
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CXA 101/Tazobactam and Metronidazole | Meropenem With Matching Saline Placebo
Number analyzed (Participants) | 61 | 25
percentage of subjects | 83.6 [71.9 to 91.8] | 96.0 [79.6 to 99.9]
Statistical Analysis 1: Comparison: CXA 101/Tazobactam and Metronidazole vs Meropenem With Matching Saline Placebo; Test type: Superiority or Other; Risk Difference (RD) = -12.4

2. Secondary Outcome: Microbiological Response of CXA 101/Tazobactam and Metronidazole at the TOC Visit in the Microbiologically Evaluable (ME) Population
Description: Microbiological response is eradication (absence of the baseline pathogen from a suitable intra-abdominal specimen) or presumed eradication (absence of a suitable intra-abdominal specimen to culture at the TOC visit in a subject who is assessed as a clinical cure at TOC)
Time Frame: Test-of-Cure Visit (7-14 days after EOT)
Population: Microbiologically Evaluable: treated subjects, with baseline pathogen susceptible to study drug, complied with protocol
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CXA 101/Tazobactam and Metronidazole | Meropenem With Matching Saline Placebo
Number analyzed (Participants) | 53 | 24
percentage of subjects | 90.6 [79.3 to 96.9] | 95.8 [78.9 to 99.9]
Statistical Analysis 1: Comparison: CXA 101/Tazobactam and Metronidazole vs Meropenem With Matching Saline Placebo; Test type: Superiority or Other; Risk Difference (RD) = -5.2

ADVERSE EVENTS:
Arm/Group | CXA 101/Tazobactam and Metronidazole | Meropenem With Matching Saline Placebo
Serious Adverse Events (participants affected / at risk) | 14/82 | 2/39
Other Adverse Events (participants affected / at risk) | 30/82 | 12/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CXA 101/Tazobactam and Metronidazole (N=82) | Meropenem With Matching Saline Placebo (N=39)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CXA 101/Tazobactam and Metronidazole (N=82) | Meropenem With Matching Saline Placebo (N=39)
Nausea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Ileus (Gastrointestinal disorders) | 3 | 0
Pyrexia (General disorders) | 12 | 4
Hypertension (Vascular disorders) | 4 | 2
Phlebitis (Vascular disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Authorship on any primary publication of the results from this study will be based on contributions to study design, enrollment, data analysis, and interpretation of results. All investigators who enroll at least one subject will be acknowledged in any journal publication.